CLINICAL TRIAL: NCT06559995
Title: Effects of Ketone Supplementation on Alcohol Withdrawal and Brain Metabolism in Alcohol Use Disorder
Acronym: KSAW
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 856689; 5R21AA031337 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-08-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder; Alcohol Withdrawal; Ketosis
Keywords: Alcohol Use Disorder; Alcohol Withdrawal; ketosis; Ketone Supplement
MeSH Terms: conditions — Alcoholism; Ketosis | interventions — Ketones

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-groups design clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone Supplement (Experimental): Ketone supplement "D-beta-hydroxybutryric acid and R-1,3 butanediol" (Kenetik: Ketone Drink, VitaNav Inc., Washington D.C.) 12g of ketones, three times a day before meals, by mouth for 4 days plus 1 dose on day 5 for magnetic resonance imaging session visit.
  Interventions: Dietary Supplement: ketone supplement "D-beta-hydroxybutryric acid and R-1,3 butanediol" 12g of ketones,; Diagnostic Test: magnetic resonance imaging session
- Placebo Beverage (Placebo Comparator): Placebo beverage, visually matched, three times a day before meals, by mouth for 4 days plus 1 dose on day 5 for magnetic resonance imaging session visit.
  Interventions: Diagnostic Test: magnetic resonance imaging session; Dietary Supplement: Placebo beverage

INTERVENTIONS:
Dietary Supplement: ketone supplement "D-beta-hydroxybutryric acid and R-1,3 butanediol" 12g of ketones, — ketone supplement
  Other Names: Kenetik: Ketone Drink, VitaNav Inc., Washington D.C.
  Arms: Ketone Supplement
Diagnostic Test: magnetic resonance imaging session — 1.5 hour magnetic resonance imaging session
  Other Names: MRI
Dietary Supplement: Placebo beverage — Placebo beverage, visually matched, three times a day before meals, by mouth for 4 days plus 1 dose on day 5 for magnetic resonance imaging session visit.
  Other Names: Placebo
  Arms: Placebo Beverage

SUMMARY:
The goal of this clinical trial is to learn the effects of ketone supplement compared to placebo on alcohol withdrawal symptoms during a 4 day alcohol withdrawal management treatment in adults with moderate to severe alcohol use disorder at the Hospital of the University of Pennsylvania, Cedar Detox Center.

DETAILED DESCRIPTION:
This is a 4-day randomized double-blinded intervention study of 30 treatment seeking adults with alcohol use disorder, who are receiving alcohol detoxification treatment at the Hospital of the University of Pennsylvania, Cedar Detox Center. Within 24 hours of admission to the inpatient unit, participants will be consented and randomized to receive 3x daily of 12g of KS (n=15; 1,3-butanediol and D-hydroxybutyric acid from Kenetik, VitaNav Inc., Washington D.C.) for 4 days or placebo beverage (n=15). Benzodiazepines and other "comfort" medications will be administered daily following the HUP Cedar withdrawal management protocol, with benzodiazepines administered based on withdrawal symptoms, monitored with the revised Clinical Institute Withdrawal Assessment for Alcohol. The revised Clinical Institute Withdrawal Assessment for Alcohol is given three or more times a day clinically to determine patient withdrawal levels and adjust medication dosages. Total daily maximum revised Clinical Institute Withdrawal Assessment for Alcohol scores, benzodiazepine dosage, and other "comfort" medications will be analyzed with a repeated measures design, with a binary factor for intervention, factor of time, and intervention by time interaction. Daily mood questions and alcohol craving questions will assess differences between treatment groups. After 4 days of study intervention, all participants will undergo an approximately 1.5-hr. magnetic resonance imaging session.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate English and provide written informed consent
2. Meets current DSM-5 criteria for moderate or severe AUD and seeking treatment for AUD
3. Minimum 3-year history of heavy drinking (self-report).
4. Presence of alcohol withdrawal (DSM-5)

Exclusion Criteria:

1. Current DSM-5 diagnosis of a major psychiatric disorder (other than alcohol and nicotine use disorders) that would interfere with study procedures.
2. Major medical problems that could impact brain function or the use of a Ketone supplement (e.g., epilepsy or diabetes) as determined by history and physical exam.
3. Clinically significant laboratory findings that could affect brain function (e.g., HIV+)
4. Head trauma with loss of consciousness for more than 30 minutes,
5. Pregnant or breast-feeding
6. BMI greater than 35
7. Self-reported claustrophobia
8. Contraindications to MRI (e.g., metal in the body that cannot be removed).
9. Current, gastrointestinal (GI), liver or other clinically significant physical disease that may interfere with the intake of the Ketone Supplement based on medical history, and evaluation of the Study Physician.
10. Current significant withdrawal from other substances, including benzodiazepines, opioids that require medication management for withdrawal and may interfere with study results/withdrawal management plan.
11. Judged by the principal investigator, Study Physician, or their designee to be an unsuitable candidate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Group changes in the total milligrams of benzodiazepines given to subjects during alcohol withdrawal management after receiving either ketone supplement or placebo beverage after 4 days of study intervention. | 4 days
  Patients in alcohol withdrawal management receive benzodiazepines measured in milligrams to treat their alcohol withdrawal symptoms. The primary outcome of this study is to compare the group differences in the amounts of benzodiazepines given to subjects after receiving either a ketone supplement or placebo beverage after 4 days, while undergoing in-patient acute withdrawal management.

SECONDARY OUTCOMES:
To measure the group differences of BHB levels in millimoles, in subjects receiving ketone supplement, Kenetik three times daily, versus a placebo beverage after 4 days of study intervention. | 4 days
  Subjects will undergo a high-field strength, 7 Tesla 1H-MRS scan to measure brain BHB levels in millimoles after the 4 days of the study intervention.
To measure the group differences of Gamma-Aminobutyric Acid levels in millimoles in subjects receiving a ketone supplement, Kenetik three times daily, versus a placebo beverage after 4 days of study intervention. | 4 days
  Subjects will undergo a high-field strength, 7 Tesla 1H-MRS scan to measure brain Gamma-Aminobutyric Acid levels in millimoles after the 4 days of the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Corinde Wiers, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Studies of Addiction, Philadelphia, Pennsylvania, United States